CLINICAL TRIAL: NCT01661491
Title: Microbiome Acquisition and Progression of Inflammation and Airway Disease in Infants and Children With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1206010476
Record Dates: First submitted 2012-08-06; First posted 2012-08-09 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fecal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cystic Fibrosis: Infants and toddlers with Cystic Fibrosis
- Non-cystic fibrosis controls: Infants and toddlers without Cystic Fibrosis

SUMMARY:
Cystic Fibrosis (CF) is a fatal, recessive genetic disorder characterized by progressive inflammation and lung damage. It is unclear whether current treatment strategies, which focus on detection and eradication of pathogenic microorganisms in the lung, are the best way to prevent the initiation of early inflammation and lung damage. This study asks how early acquisition of microbial flora occurs in infants with CF and healthy baby controls, and whether this process initiates or influences early inflammation and clinical disease progression in CF.

DETAILED DESCRIPTION:
Cystic Fibrosis is the most common lethal genetic disorder in Caucasian populations. Mutations of the Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) affect its ability to act as a chloride channel. The recent development of a transgenic pig model of CF has demonstrated that newborn CF lungs, free of bacteria and inflammation at birth, become colonized with a mixed microbial flora that likely initiates early inflammatory changes which precede clinically apparent deterioration in lung function.

Because chronic infection and inflammation play central roles in CF disease progression and exacerbations, many clinicians and researchers have focused on identifying pathogens associated with CF infection and inflammation. Recent studies outside the area of CF, however, have clearly demonstrated that "non-pathogens", such as the commensal flora carried by all humans at multiple mucosal sites, engage the host's innate and adaptive immune systems constantly. This interaction between "microbiome" and host genome is responsible for appropriate development and function of protective inflammatory and immune responses.

We hypothesize that acquisition of a commensal flora by newborns with CF may play a critical role in initiating pathogenic inflammatory responses that subsequently lead to lung damage. The acquired commensal flora may initially be identical to that of a non-CF infant, but may be altered by the direct or indirect effects of CFTR mutation on the mucosal environment. Such an altered flora is likely to encode different metabolic and regulatory functions, and may directly influence host inflammatory responses. If so, a novel therapeutic opportunity may exist to modulate this commensal flora, or to manipulate its immunomodulatory functions in a way that interrupts the insidious cycle of inflammation and damage that characterizes CF.

We propose to test our hypothesis in three specific aims: (1) Describe the acquisition and evolution of gut and respiratory tract microbiomes in CF infants and non-CF controls; (2) Determine the relationship between the microbiota and markers of inflammation in these two cohorts; and (3) Determine whether early declines in lung function are associated with inflammatory biomarkers or microbiome composition/function. This study is novel in its focus on a rarely studied population, at a time when interventions might significantly impact progression of this lethal disease and preserve pulmonary function. Its innovation lies in applying state of the art technologies and methods to samples that can be collected simply and non-invasively, thus increasing the likelihood that the findings of this study can be translated into clinical practice.

ELIGIBILITY:
Cystic Fibrosis participants:

Inclusion Criteria:

* laboratory diagnosis of Cystic Fibrosis

Exclusion Criteria:

* Major organ system disease other than Cystic Fibrosis
* History of prematurity

Non Cystic Fibrosis control participants:

Inclusion Criteria:

* Proof of a negative newborn CF screening test

Exclusion Criteria:

* Major organ system disease
* History of prematurity

Ages: 3 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants and children up to the age of 4 with Cystic Fibrosis, and age-matched controls without cystic fibrosis will be eligible for this study. Participants will be recruited from the Cystic Fibrosis clinic and Primary Care Clinic of the Yale New Haven Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Average Unifrac Value in Fecal Microbiome & Metagenome Composition at 4 years | 4 years
  High throughput sequencing will be used to identify microbial taxa and microbial genes present in feces, and to determine how these change over a period of 4 years

SECONDARY OUTCOMES:
Change from Baseline in the Amounts of Calprotectin at 4 years | 4 years
  Fecal calprotectin will be measured by elisa
Change from Baseline in the Amounts of Short Chain Fatty Acids at 4 years | 4 years
  Fecal short chain fatty acids will be measured by gas chromatography

CONTACTS AND LOCATIONS:
Overall Officials: Barbara I Kazmierczak, MD PhD, Principal Investigator — Yale University; Marie Egan, MD, Principal Investigator — Yale University
Locations (1):
- Cystic Fibrosis Clinic, Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No